CLINICAL TRIAL: NCT05568550
Title: Phase II Study of Pembrolizumab in Combination With Radiation With or Without Olaparib in Localized High-risk Prostate Cancer
Brief Title: Pembro With Radiation With or Without Olaparib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zin W Myint (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Zin W Myint, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22-GU-80
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: immunotherapy; PARP; radiation; androgen deprivation therapy; ADT; PD-1
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab; olaparib; Androgen Antagonists; Radiotherapy

STUDY DESIGN:
Intervention Model Description: 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 - Pembrolizumab and Olaparib (Experimental): Patients with high-risk prostate cancer receiving combination therapy with Pembrolizumab and Olaparib.
  Interventions: Biological: Pembrolizumab; Drug: Olaparib; Drug: Androgen Deprivation Therapy; Radiation: Radiation Therapy
- Arm 2 - Pembrolizumab (Experimental): Patients with high-risk prostate cancer receiving combination therapy with Pembrolizumab.
  Interventions: Biological: Pembrolizumab; Drug: Androgen Deprivation Therapy; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab will be delivered via IV at 200mg on day 1 of each 3-week cycle for approximately 12 months. Cycle 1 begins 21 days prior to radiation therapy and cycles 2-17 are administered during and after radiation therapy.
  Other Names: Keytruda
Drug: Olaparib — 200mg Olaparib will be given twice daily for a total of 3 cycles. Cycle 1 begins 21-days prior to radiation therapy.
  Other Names: Lynparza
  Arms: Arm 1 - Pembrolizumab and Olaparib
Drug: Androgen Deprivation Therapy — Androgen Deprivation Therapy (either LHRH agonist or LHRH antagonist) as per treating physician choice will be allowed within 3 months prior to randomization. Duration is per institutional standards.
Radiation: Radiation Therapy — Definitive radiation (total dose and fractions) will be dosed per institutional standards. Definitive radiation may include external beam radiation therapy with or without brachytherapy, based on NCCN risk score and as per treating physicians.

SUMMARY:
This trial will evaluate whether the immune-sensitizing effects of immunotherapy (Pembrolizumab) and radiation with or without a PARP-inhibitor (Olaparib) will increase the effects of immunotherapy in men with high-risk localized prostate cancer.

DETAILED DESCRIPTION:
Immunotherapy and PARP-inhibitor are known to have radio-sensitizing effects when combined with radiation therapy. In addition, the combination with PARP-inhibitor and radiation can increase neoantigen expression, cytotoxic lymphocyte infiltration within the tumor microenvironment and increased immune stimulating cytokine concentration. Thus, there is a potential synergy of combining immunotherapy and PARP-inhibitor.

This is a phase 2 randomized 1:1 study. Subjects will be randomized to one arm (pembro + PARPi + standard of care therapy which is definitive radiation therapy combined with hormonal therapy) vs. another arm (pembro + standard of care therapy). All subjects will receive adjuvant immunotherapy for one year once they are done with definitive radiation treatment.

Due to slow accrual and feasibility concerns, the protocol was modified to single arm phase II study. All patients will receive definitive radiation therapy combined with ADT per institutional standards. In addition to concurrent ADT and radiation therapy, patients on this trial will also receive as follow: Pembrolizumab (17 cycles) combined with olaparib (the first three cycles). The remaining patients will be enrolled to Arm 1 only (i.e., Arm 2 usual care is closed to accrual upon Amendment 5 protocol).

ELIGIBILITY:
Inclusion Criteria:

* Male participants with histologically confirmed adenocarcinoma of the prostate
* High-risk / very high-risk status per NCCN guidelines
* ECOG performance status 0 to 1
* Regional lymph nodes are allowed.
* Agree to use contraception during the treatment period and for at least 120 days after the last dose of study intervention and refrain from donating sperm during this period.
* Ability to understand and the willingness to sign a written informed consent document.
* Adequate organ and marrow function
* Prior pharmacologic androgen ablation for prostate cancer is allowed only if the onset of androgen ablation is ≤90 days prior to the date of registration
* Known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.

Exclusion Criteria:

* Prior hormonal therapy with LHRH agonists (e.g., Lupron) and LHRH antagonists (e.g., Degarelix)for prostate cancer continuously for more than 90-days prior to study enrollment.
* Prior radiation to the prostate or pelvic nodes radiation.
* Previous or major surgery (colorectal anastomosis, total cystectomy, etc.).
* History of Ulcerative proctitis.
* Concurrent active, additional malignancy in the last 2 years.
* Prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization.
* Patients with M1 disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2029-07-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Response Rate | 6 months
  The proportion of patients who achieve a PSA nadir level of ≤ 0.06ng/mL six months after completion of radiation therapy.

SECONDARY OUTCOMES:
Biochemical-Free Survival | 3 years
  Biochemical-free survival rate at 3 years as defined by Phoenix Criteria.
Metastasis-Free Survival | 3 years
  Metastasis-free survival rate at 3 years as defined by RECIST v1.1 criteria.
Time to Normalization of Serum Testosterone | 3 years
  Time from normalization is the date of first return to normal serum testosterone 270 ng/ml or greater after withdrawal of androgen deprivation therapy.
Molecular Alterations in Homologous Recombination Repair Genes | 3 years
  Molecular alterations in the homologous recombination repair (HHR) genes.

OTHER OUTCOMES:
PSA Progression-Free Survival | 3 years (Pre-treatment baseline, cycle 3, 6 months or at disease progression)
  PSA progression-free survival (PSA-PFS) stratified by PDL1 immunohistochemistry expression on baseline or /archival biopsy tissue, if tissue is available.
Correlation between clinical outcome and immune cell subtype. | 3 years (Pre-treatment baseline, cycle 3, 6 months or at disease progression)
  Correlation between the clinical outcomes and changes in immune cell subtype frequencies (% CD4 T cells, % CD8 T cells, % naïve, effector memory, and T regulatory cells) immune functions (T cell ability to induce cytokine following stimulation).
Correlation between clinical outcome and cytokine levels. | 3 years (Pre-treatment baseline, cycle 3, 6 months or at disease progression)
  Correlation between the serum cytokines (IL2, IL-10, and INF-γ) and clinical outcomes.
Correlation between clinical outcomes and TCR repertories clonotypes. | 3 years (Pre-treatment baseline, cycle 3, 6 months or at disease progression)
  Correlation between T cell receptor (TCR) repertories clonotypes and clinical outcomes.
Percent changes in plasma circulating tumor DNA | Baseline and on-treatment (6 months)
  Percent changes in plasma circulating tumor DNA (ctDNA).

CONTACTS AND LOCATIONS:
Overall Officials: Zin W Myint, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No